CLINICAL TRIAL: NCT01951378
Title: Comparison of a Breath Enhanced High Density Jet Nebulizer With a Standard Jet Nebulizer for the Treatment of Children With a Moderate to Severe Asthma Exacerbation in the Emergency Department
Brief Title: Comparison of Nebulizers in ED in Pediatric Asthma Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No data are available for this study as the PI has left the institution.
Sponsor: Seton Healthcare Family (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CR-13-119
Record Dates: First submitted 2013-09-04; First posted 2013-09-26 (Estimated); Results first posted 2020-09-02 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2020-08

CONDITIONS: Asthma
Keywords: Asthma; Asthma exacerbation
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hudson RCI® nebulizer (Active Comparator): Patients randomized to the "standard" arm will receive treatments as dictated by our standard ED asthma pathway (Fig. 1). All treatments will be administered with our standard ED nebulizer, the Hudson RCI® Up-Draft® Neb-U-Mist® nebulizer (Teleflex Medical®, Research Triangle Park, NJ), and a simple mask (Hudson RCI®, Teleflex Medical®, Research Triangle Park, NJ).
  Interventions: Device: Hudson RCI® nebulizer; Drug: Albuterol
- NebuTech® HDN® nebulizer (Active Comparator): Patients randomized to the "NebuTech®" arm will receive treatments as dictated by our trial pathway, referred to as the "rapid Albuterol/Proventil delivery pathway" (Fig. 2). All nebulizations in this arm will be administered via the Breath-Enhanced High Density Jet Nebulizer, NebuTech® HighDensityNebulizer®,(Salter Labs®, Arvin, CA). Respiratory Therapists (RT) will attempt to deliver all treatments with a mouthpiece, as that has been shown to be the most efficient and reliable mode of aerosol delivery for most children 31, 32. If the Respiratory Therapist feels that the child will not or cannot effectively use a mouthpiece, a mask will be used.
  Interventions: Device: NebuTech® HDN® nebulizer; Drug: Albuterol

INTERVENTIONS:
Device: Hudson RCI® nebulizer — After the first hour of treatment, patients in the standard arm will receive a repeat assessment, including all of the measurements collected at baseline as well as reported side effects. Those patients who score PAS 0-2 will then be discharged home, after an optional observation period, as per the pathway. Those who score PAS > 2 will receive a second treatment. At the end of the second treatment patients will again be re-assessed, and repeat measurements obtained. At that time, depending on the patient's PAS score, he/she will be dispositioned to home, the floor, the pulmonary high acuity unit (PHAU), or the pediatric intensive care unit (PICU).
  Arms: Hudson RCI® nebulizer
Device: NebuTech® HDN® nebulizer — All treatments in the NebuTech® arm will be given at a standard dilution of 5 ml (diluted with normal saline to a total volume of 5 ml as per the manufacturer's recommendation). Patients in this arm will receive up to four treatments with parameters measured after each treatment, similar to the control arm. Patients who complete four treatments will then be dispositioned based on PAS score, similar to the control arm. Subjects may have started treatment prior to consent and may receives unit dose (2.5 mg) Albuterol/Proventil treatments will be given with a standard nebulizer up to 3 times as needed and may change over to study randomized device once consented to eith arm.
  Arms: NebuTech® HDN® nebulizer
Drug: Albuterol — Subjects may have started treatment prior to consent and may receives unit dose (2.5 mg) Albuterol/Proventil treatments will be given with a standard nebulizer up to 3 times as needed and may change over to study randomized device once consented to eith arm.
  Other Names: Proventil

SUMMARY:
The primary objective will be, in an open-label randomized trial, a comparison of emergency department (ED) length of stay (LOS) between children experiencing acute asthma treated with two different nebulizers. Secondary outcomes will include admission rates, hospital LOS, need for additional therapies, transfers to a higher level of care, side-effects, and unscheduled return visits

DETAILED DESCRIPTION:
To our knowledge, no study has compared a breath-enhanced nebulizer to a standard jet nebulizer for the treatment of acute asthma in children. The goal of this study is to determine whether a rapid albuterol delivery pathway with a breath-enhanced nebulizer can reduce ED LOS, while maintaining admission rates, repeat visits, adjunctive therapies, and side-effects, when compared to a traditional asthma pathway with a standard jet nebulizer. The Salter® Nebutech® HDN® was chosen because its breath-enhanced design and bolus delivery system may deliver greater amounts of albuterol to the small airways, in a shorter period of time, when compared with standard jet nebulizers and other nebulizers in its class.

The study site will be a large, urban pediatric emergency department (ED) with approximately 80,000 visits per year. The study protocol will be submitted to the hospital's Institutional Review Board (IRB) for approval. Children will be eligible for enrolment if they are between 3 and 18 years of age and present to the ED with an acute asthma exacerbation of at least moderate severity. The lower age cutoff was chosen because asthma diagnosis and beta agonist response can be unreliable in younger children. The upper age cutoff was chosen to include only pediatric patients, as this is a pediatric asthma study. Children must have a history of physician-diagnosed asthma as reported by the parent or guardian. Children will be enrolled when a research team member is available to obtain informed consent (convenience sample). Children will be excluded from enrollment if the initial pediatric asthma score (PAS) is < 3, immediate resuscitation is required, they have a history of chronic lung disease or congenital heart disease, they have any neuromuscular disease, intrathoracic foreign body is suspected, they are or may be pregnant, they are currently breast feeding, they have received oral or parenteral steroids within the last week (inhaled steroids are allowed), or they have an allergy or other contraindication to one of the study medications.

Potential subjects will be identified in triage and screened for enrolment if study personnel are available. If consented, the patient will be randomized to one of the two treatment arms. If there will be greater than a 15 minute delay in treatment due to the consent process, unit dose (2.5 mg) albuterol treatments will be given with a standard nebulizer up to 3 times as needed. That patient may still be enrolled provided he/she still meets inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 3 years and < 18 years
* History of physician-diagnosed asthma
* Presenting to ED with acute asthma exacerbation according to attending physician

Exclusion Criteria:

* PAS score < 3
* Immediate resuscitation required
* Chronic lung disease (other than asthma)
* Congenital heart disease 5. Neuromuscular disease 6. Suspected intrathoracic foreign body 7. Is or may be pregnant 8. Currently breast feeding 9. Oral or parenteral steroids within the last 7 days 10. Allergy or other contraindication to any of the study medications

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew H. Wilkinson, MD, Principal Investigator — Seton Healthcare Family
Locations (1):
- Dell Children's Medical Center of Central Texas, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Hudson RCI® Nebulizer: Patients randomized to the standard arm will receive treatments as dictated by our standard ED asthma pathway (Fig. 1). All treatments will be administered with our standard ED nebulizer, the Hudson RCI® Up-Draft® Neb-U-Mist® nebulizer (Teleflex Medical®, Research Triangle Park, NJ), and a simple mask (Hudson RCI®, Teleflex Medical®, Research Triangle Park, NJ).
  Hudson RCI® nebulizer: After the first hour of treatment, patients in the standard arm will receive a repeat assessment, including all of the measurements collected at baseline as well as reported side effects. Those patients who score PAS 0-2 will then be discharged home, after an optional observation period, as per the pathway. Those who score PAS > 2 will receive a second treatment. At the end of the second treatment patients will again be re-assessed, and repeat measurements obtained. At that time, depending on the patient's PAS score, he/she will be dispositioned to home, the floor, the pulmonary high acuity unit (PHA
- NebuTech® HDN® Nebulizer: Patients randomized to the NebuTech® arm will receive treatments as dictated by our trial pathway, referred to as the "rapid Albuterol/Proventil delivery pathway" (Fig. 2). All nebulizations in this arm will be administered via the Breath-Enhanced High Density Jet Nebulizer, NebuTech® HighDensityNebulizer®,(Salter Labs®, Arvin, CA). Respiratory Therapists (RT) will attempt to deliver all treatments with a mouthpiece, as that has been shown to be the most efficient and reliable mode of aerosol delivery for most children 31, 32. If the Respiratory Therapist feels that the child will not or cannot effectively use a mouthpiece, a mask will be used.
  NebuTech® HDN® nebulizer: All treatments in the NebuTech® arm will be given at a standard dilution of 5 ml (diluted with normal saline to a total volume of 5 ml as per the manufacturer's recommendation). Patients in this arm will receive up to four treatments with parameters measured after each treatment, similar to the control arm. Patient
Period: Overall Study
Arm/Group | Hudson RCI® Nebulizer | NebuTech® HDN® Nebulizer
Started | 23 | 17
Completed | 0 | 0
Not Completed | 23 | 17
Not completed — Study Terminated-Not completed | 23 | 17

BASELINE CHARACTERISTICS:
Groups:
- Hudson RCI® Nebulizer: Patients randomized to standard arm receives treatments per standard ED asthma pathway. Treatments administered with standard ED nebulizer, Hudson RCI® Up-Draft® Neb-U-Mist® nebulizer (Teleflex Medical®, Research Triangle Park, NJ), and a simple mask (Hudson RCI®, Teleflex Medical®, Research Triangle Park, NJ).
  Hudson RCI® nebulizer: After 1 hour, patients in standard arm receive another assessment, with all baseline measurements and reported side effects. Patients who score PAS 0-2 will be discharged, after optional observation period, per pathway. Those who score PAS > 2 receive second treatment, then re-assessed, and measurements repeated. Then, depending on PAS score, he/she will be sent, the floor, the pulmonary high acuity unit (PHAU), or PICU.
  Albuterol: Subjects may begin treatment before consent and may receive 2.5 mg Albuterol/Proventil treatments given with standard nebulizer <3 times as needed and may change over to study randomized device once consented to either arm.
- NebuTech® HDN® Nebulizer: Randomized patients receive treatments per "rapid Albuterol/Proventil delivery pathway". Nebulizations given via Breath-Enhanced High Density Jet Nebulizer, NebuTech® HighDensityNebulizer®,(Salter Labs®, Arvin, CA). If child will not or cannot use mouthpiece, a mask will be used.
  NebuTech® HDN® nebulizer: Treatments are dilution of 5 ml. Patients receive <4 treatments with measurements after each. Patients who complete 4 treatments will be dispositioned based on PAS score. Subjects may begin treatment before consent and may receive 2.5 mg Albuterol/Proventil treatments via standard nebulizer <3 times as needed and may change to study randomized device once consented to either arm.
  Albuterol: Subjects may start treatment before consent and may receives 2.5 mg Albuterol/Proventil given with standard nebulizer <3 times as needed and may change over to study randomized device once consented to either arm.
- Total: Total of all reporting groups
Arm/Group | Hudson RCI® Nebulizer | NebuTech® HDN® Nebulizer | Total
Number analyzed (Participants) | 23 | 17 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 17 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11 (5) | 9 (5) | 10 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 13 | 11 | 24
Region of Enrollment [Number; unit: participants]
  United States | 23 | 17 | 40

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective Will be, in an Open-label Randomized Trial, a Comparison of Emergency Department (ED) Length of Stay (LOS) Between Children Experiencing Acute Asthma Treated With Two Different Nebulizers
Description: The primary endpoint will be mean ED LOS difference between the groups. Using historical data as a guide, we calculated a baseline LOS mean for discharged patients of 181 minutes, and standard deviation (SD) of 83 minutes. For this reason, an interim analysis will be conducted in order to assess a pilot sample for the purpose of estimating these values. 25 subjects in each arm (50 subjects total) will be enrolled during the initial phase of the study. This early phase interim analysis is not powered to test for differences between the groups, but establish pilot-phase findings that can be used for more accurate sample size calculation. However, the primary outcome of ED LOS will then be tested to determine the difference between study arms, using the non-parametric Mann-Whitney U test due to the likely skewed-nature of the distribution of ED LOS values for the purpose of establishing an estimate of effect size in the initial enrollment phase.
Time Frame: 1 year
Population: No data are available for this study as the PI has left the institution and no study team member is present. The local IRB closed and was replaced in July 2017 by the University of Texas. Sincere efforts were made to obtain the data for reporting, however, no data are available
Groups:
- Hudson RCI® Nebulizer: Patients randomized to "standard" arm receives treatments by standard ED asthma pathway. Treatments administered with standard ED nebulizer, Hudson RCI® Up-Draft® Neb-U-Mist® nebulizer (Teleflex Medical®, Research Triangle Park, NJ), and simple mask (Hudson RCI®, Teleflex Medical®, Research Triangle Park, NJ). Hudson RCI® nebulizer: After 1 hour, patients in standard arm have repeat assessment, with all measurements collected at baseline and reported side effects. Patients who score PAS 0-2 will be discharged after observation, per pathway. Those who score PAS > 2 receive second treatment. After second treatment patients re-assessed, and repeat measurements obtained. Then, based on score, he/she will be dispositioned home, the floor, pulmonary high acuity unit (PHAU), or (PICU).
  Albuterol: Subjects may have treatment before consent and may receive 2.5 mg treatments with standard nebulizer up to 3 times as needed and may change to randomized device once consented to either arm.
- NebuTech® HDN® Nebulizer: Patients randomized to "NebuTech®" arm receive treatments by, "rapid Albuterol/Proventil delivery pathway", given by Breath-Enhanced High Density Jet Nebulizer, NebuTech® HighDensityNebulizer®,(Salter Labs®, Arvin, CA). Respiratory Therapists (RT) will try to give treatments with mouthpiece, shown most efficient and reliable mode of aerosol delivery for children. If RT feels child will not or cannot use a mouthpiece, a mask will be used.
  NebuTech® HDN® nebulizer: Treatments given at 5 ml (diluted with normal saline). Patients complete <4 treatments, dispositioned based on PAS. Subjects may start treatment before consent and may receive 2.5 mg Albuterol/Proventil treatments given with standard nebulizer <3 times as needed and may change to study randomized device once consented.
  Albuterol: Subjects start treatment before consent and may receive 2.5 mg. Treatments receive standard nebulizer up to 3 times as needed and may change to randomized device once consented to either arm.
Arm/Group | Hudson RCI® Nebulizer | NebuTech® HDN® Nebulizer
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: to Evaluate Admission Rates.
Description: Baseline characteristics (demographics, history, and clinical characteristics of presentation) of subjects in each treatment arm will be summarized in a table. These descriptive characteristics will be compared between arms using standard t-test or a non-parametric alternative for linear values (eg, age) and chi-squared tests for binomial or categorical values (eg, gender) with p-values reported in the summary table.
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | Hudson RCI® Nebulizer | NebuTech® HDN® Nebulizer
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Will Evaluate Hospital LOS. Safety Issue?: (FDAAA) No
Description: as for outcome 2
Time Frame: 1 year
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Will Evaluate Need for Additional Therapies.
Description: as for outcome 2
Time Frame: 1 year
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Will Evaluate Transfers to a Higher Level of Care.
Description: as for outcome 2
Time Frame: 1 year
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Will Evaluate for Unscheduled Return Visits.
Description: as for outcome 2
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: No data are available for this study as the PI has left the institution and no study team member is present. The local IRB closed and was replaced in July 2017 by the University of Texas. Sincere efforts were made to obtain the data for reporting, however, no data are available
Description: No data are available for this study as the PI has left the institution and no study team member is present. The local IRB closed and was replaced in July 2017 by the University of Texas. Sincere efforts were made to obtain the data for reporting, however, no data are available
Groups:
- Hudson RCI® Nebulizer: Patients randomized to standard arm receive treatments by standard ED asthma pathway. Treatments administered with standard ED nebulizer, the Hudson RCI® Up-Draft® Neb-U-Mist® nebulizer (Teleflex Medical®, Research Triangle Park, NJ), and a simple mask (Hudson RCI®, Teleflex Medical®, Research Triangle Park, NJ).
  Hudson RCI® nebulizer: After 1 hour, patients in standard arm receive repeat assessment, including baseline measurements and reported side effects. Patients who score PAS 0-2 sent home, after optional observation period, per pathway. Those with score PAS > 2 receive second treatment, re-assessed, and repeat measurements. Based on patient's PAS score, he/she will be dispositioned home, the floor, the pulmonary high acuity unit (PHAU), or the pediatric intensive care unit (PICU).
  Albuterol: Subjects may start treatment before consent and receive 2.5 mg. Albuterol/Proventil treatments by standard nebulizer <3 times as needed and may change to study randomized device once c
- NebuTech® HDN® Nebulizer: Patients randomized to "NebuTech®" arm will receive treatments as dictated by our trial pathway, referred to as the "rapid Albuterol/Proventil delivery pathway" (Fig. 2). All nebulizations in this arm will be administered via the Breath-Enhanced High Density Jet Nebulizer, NebuTech® HighDensityNebulizer®,(Salter Labs®, Arvin, CA). Respiratory Therapists (RT) will attempt to deliver all treatments with a mouthpiece, as that has been shown to be the most efficient and reliable mode of aerosol delivery for most children 31, 32. If the Respiratory Therapist feels that the child will not or cannot effectively use a mouthpiece, a mask will be used.
  NebuTech® HDN® nebulizer: All treatments in the NebuTech® arm will be given at a standard dilution of 5 ml (diluted with normal saline to a total volume of 5 ml as per the manufacturer's recommendation). Patients in this arm will receive up to four treatments with parameters measured after each treatment, similar to the control arm. Patient
Arm/Group | Hudson RCI® Nebulizer | NebuTech® HDN® Nebulizer
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No